CLINICAL TRIAL: NCT02919020
Title: Efficacy of Proprioceptive Neuromuscular Facilitation About Functional Performance, Pain and Quality of Life in Older Women With Gonarthrosis: Randomized Controlled Trial
Brief Title: Efficacy of Proprioceptive Neuromuscular Facilitation in Older Women With Gonarthrosis
Acronym: PNF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Collaborators: Daniella Araújo de Oliveira (Unknown); Angélica da Silva Tenório (Unknown)
Responsible Party: Principal Investigator, Thaís Ferreira Lopes Diniz Maia, Investigador Principal, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ECR2015
Record Dates: First submitted 2016-09-24; First posted 2016-09-29 (Estimated); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Osteoarthritis Knee
Keywords: Proprioceptive Neuromuscular Facilitation (PNF ); resistance exercise
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Muscle Stretching Exercises; Resistance Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Proprioceptive neuromuscular facilitation (PNF); (Experimental): Proprioceptive neuromuscular facilitation, using the technique of rhythmic initiation and Combination of Isotonic on lower members
  Interventions: Other: Proprioceptive neuromuscular facilitation (PNF)
- resistance exercise (Experimental): Resistance exercise to strengthen lower limbs
  Interventions: Other: Resistance exercise

INTERVENTIONS:
Other: Proprioceptive neuromuscular facilitation (PNF) — Proprioceptive neuromuscular facilitation, using the technique of rhythmic initiation and Combination of Isotonic on lower members
  Arms: Proprioceptive neuromuscular facilitation (PNF);
Other: Resistance exercise — resistance exercise to strengthen lower limbs
  Arms: resistance exercise

SUMMARY:
To evaluate the effectiveness of the method Proprioceptive Neuromuscular Facilitation (PNF) as physical therapy approach to the reduction of pain and improvement in functional performance and quality of life in women with knee osteoarthritis.

DETAILED DESCRIPTION:
Patients will be divided into two groups: group perform proprioceptive neuromuscular facilitation and other group submit performing resistance exercises.

ELIGIBILITY:
Inclusion Criteria:

* Women;
* Age between 50 and 80 years;
* Clinical diagnosis of Osteoarthritis of knees ;
* Patients with presence of at least 90 ° range of motion of knee flexion ;
* Do not practitioners of physical exercise and physical therapy during the period of participation in the survey

Exclusion Criteria:

* Diagnosis of other rheumatological and neurological diseases ;
* orthopedic surgery History in the lower limbs ;
* Individuals with muscle strength of the lower limbs <3 ;
* Cognitive impairment or neurological disease that compromises the understanding and implementation of the Protocol (Mini Mental State Examination <18 for the illiterate and <24 for others);
* Body mass index ≥ 30.0 (obesity , according to the World Health Organization ) .
* Individuals classified as physical activity level "very active" by the IPAQ (International Physical Activity Questionnaire ) .

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Change in pain | "change from baseline in pain 6th - 12th week"
  "Pain control diary"
Quality of life | change from baseline in quality of life 6th-12th week
  Western Ontario and McMaster Universities Questionaire
Functional performance | Change based on functional performance 6th - 12th week
  "30 s -chair stand test"
Quality of life | Change based on functional performance 6th - 12th week
  Medical Outcomes Study 36 - Item Short - Form Health Survey
Functional Performance | Change based on functional performance 6th - 12th week
  "Walk Test of 40 meters at a rapid pace
Functional Performance | "Walk Test of 40 meters at a rapid pace
  "Stair climb test"

SECONDARY OUTCOMES:
pain sensitivity threshold | change from baseline in pain threshold 6th-12th week pressure
  "Algometry"
Range of motion | "change from baseline in the range of knee flexion 6th-12th week"
  "Universal Goniometer"

CONTACTS AND LOCATIONS:
Overall Officials: Daniella A Oliveira, Study Director — Universidade Federal de Pernambuco
Locations (1):
- Hospital Universitário Drº Washigton Antônio de Barros, Petrolina, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No